CLINICAL TRIAL: NCT07181239
Title: A Phase III, Randomized, Open-Label, Multicenter Study Comparing CM336 Monotherapy vs. Investigators Selected Standard of Care in Participants With Relapsed or Refractory Multiple Myeloma Who Have Received ≥2 Prior Lines of Therapy
Brief Title: Study of CM336 in Relapsed or Refractory Multiple Myeloma Patients
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Keymed Biosciences Co.Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CM336-021209
Record Dates: First submitted 2025-09-12; First posted 2025-09-18 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Multiple Myeloma (MM)
MeSH Terms: conditions — Multiple Myeloma | interventions — Standard of Care

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A: CM336 (Experimental)
  Interventions: Drug: CM336 Injection
- Arm B: Standard of Care Regimens (Active Comparator)
  Interventions: Drug: Standard Of Care( SOC)

INTERVENTIONS:
Drug: CM336 Injection — Specified dose on specified days
  Arms: Arm A: CM336
Drug: Standard Of Care( SOC) — Specified dose on specified days
  Arms: Arm B: Standard of Care Regimens

SUMMARY:
The purpose of this study is to compare the efficacy between CM336 and investigator's choice Standard of Care in relapsed or refractory multiple myeloma (RRMM) patients.

ELIGIBILITY:
Inclusion Criteria:

* The subjects voluntarily sign the informed consent form (ICF) and agree to abide by the provisions of this protocol.
* Age ≥ 18 years old, gender is not limited.
* Eastern Cooperative Oncology Group performance status score (ECOG) 0-2 points.
* Patients with relapsed or refractory multiple myeloma who have received at least two lines of anti-myeloma treatment previously, and must include at least one proteasome inhibitor (PI), one immunomodulatory agent (IMiD), and one anti-Cluster of Differentiation 38(CD38) monoclonal antibody.
* The subject has evidence of disease progression or has not achieved remission after the last line of treatment, as determined by the investigator based on the International Myeloma Working Group (2016) criteria.
* The subject has measurable disease at the screening period, meeting at least one of the following criteria:

  1. Serum M protein ≥ 5 g/L;
  2. Urinary M protein ≥ 200 mg/24 h;
  3. Serum free light chain (sFLC) ≥ 100 mg/L and abnormal κ/ λ ratio.

Exclusion Criteria:

* Previous receipt of any treatment targeting B-cell maturation antigen (BCMA).
* Those who are intolerant to dexamethasone will be excluded.
* Within 3 months prior to the first administration, they have received chimeric antigen receptor T cells (CAR-T) /chimeric antigen receptor Nature killer cell (CAR-NK) therapy.
* Within 3 months prior to the first administration, they have received autologous stem cell transplantation; within 6 months prior to the first administration, they have received allogeneic stem cell transplantation (for subjects who have received allogeneic transplantation, they must have discontinued all immunosuppressants for ≥ 6 weeks and have no signs of graft-versus-host disease before being eligible for enrollment).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2027-09 (Estimated); Study Completion 2030-04 (Estimated)

PRIMARY OUTCOMES:
PFS | Up to 4 years
  The progression-free survival (PFS) evaluated by Blinded Independent Central Review (BICR)

CONTACTS AND LOCATIONS:
Overall Officials: Lugui Qiu, Principal Investigator — Chinese Academy of Medical Sciences; Gang An, Principal Investigator — Chinese Academy of Medical Sciences
Locations (1):
- Institute of Hematology & Blood Diseases Hospital, Tianjin, Tianjin Municipality, China